CLINICAL TRIAL: NCT05757531
Title: Disposition of [14C]-LY3437943 Following Subcutaneous Administration in Healthy Male Participants
Brief Title: A Study of Carbon-14-Labelled [14C] LY3437943 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18217; J1I-MC-GZBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Radioactive; ADME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [¹⁴C]-LY3437943 (Experimental): Single dose of [¹⁴C]-LY3437943 administered subcutaneously (SC).
  Interventions: Drug: [¹⁴C]-LY3437943

INTERVENTIONS:
Drug: [¹⁴C]-LY3437943 — Administered SC.

SUMMARY:
The main purpose of this study is to is to look at how much LY3437943 gets into the bloodstream and how long the body takes to get rid of it in healthy male participants. This study will involve a single dose of 14C radiolabeled LY3437943. his means that a radioactive tracer substance, C14, will be incorporated into the study drug to investigate the study drug and its breakdown products and to find out how much of these pass from blood into urine, feces and expired air.

The study will last up to approximately 15 weeks including the screening period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Have a body mass index within the range 18.5 to 32.0 kilograms per meter squared (kg/m²)
* Have clinical laboratory test results within normal reference range for the population or investigative site, or results outside the normal reference range that are judged to be not clinically significant by the investigator. Participants with dyslipidemia may be included in the study, at the discretion of the investigator, as long as they fulfill other eligibility criteria
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are willing to receive study treatment by SC injections
* Have a history of a minimum of 1 bowel movement per day
* Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Have a clinically significant abnormal blood pressure and/or pulse rate as determined by the investigator at screening or check-in
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, GI, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the IP; or of interfering with the interpretation of data
* Have evidence of significant active neuropsychiatric disease, as determined by the investigator
* Show evidence of HIV infection and/or positive HIV antibodies, hepatitis C and/or positive hepatitis C antibody, hepatitis B and/or positive hepatitis B surface antigen
* Have a history of constipation or have had acute constipation within 3 weeks prior to check-in
* Have evidence of active renal disease (eg, diabetic renal disease, polycystic kidney disease) or an estimated creatinine clearance of less than 70 mL/minute, calculated using the Chronic Kidney Disease-Epidemiology equation
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) and/or elevation in serum amylase or lipase (greater than 1.5-fold the ULN) at screening
* Have used or plan to use over-the-counter or prescription medication, and/or dietary or herbal supplements (with the exception of vitamin supplements, acetaminophen and/or thyroid replacement therapy) within 14 days or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study, including any medications that reduce GI motility, including, but not limited to, anticholinergics, antispasmodics, 5 hydroxytryptamine-3 receptor antagonists, dopamine antagonists, and opiates
* Have had exposure to significant radiation within 12 months prior to dosing (eg, serial x-ray or CT scans, barium meal, being employed in a job requiring radiation exposure monitoring)
* Have participated in any clinical trial involving a radiolabeled substance within the past 12 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3437943 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to 63 days post dose
  Urinary Excretion of LY3437943 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3437943 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to 63 days post dose
  Fecal Excretion of LY3437943 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
PK: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC (0-∞)) of Total Radioactivity and [¹⁴C]-LY3437943 | Predose up to 63 days post dose
  PK: AUC (0-∞) of Total Radioactivity and [¹⁴C]-LY3437943
PK: Maximum Concentration (Cmax) of Total Radioactivity and [¹⁴C]-LY3437943 | Predose up to 63 days post dose
  PK: Cmax of Total Radioactivity and [¹⁴C]-LY3437943
Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable) | Predose up to 63 days post dose
  Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable)
Total Number of Metabolites of LY3437943 | Predose up to 63 days post dose
  Total Number of Metabolites of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No